CLINICAL TRIAL: NCT04129268
Title: Determining the Minimum Amount of Exercise to Improve Glycaemic Control in Young and Old Overweight Males, and in Patients With Type II Diabetes
Brief Title: Determining the Minimal Amount of Exercise to Improve Glycaemic Control
Acronym: MiniEx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lancaster University (Other)
Responsible Party: Principal Investigator, Dr. Chris Gaffney, Principal Investigator and Lecturer in Sports Science, Lancaster University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 248319; 19/NW/0066 (Other: NHS REC Reference)
Record Dates: First submitted 2019-10-09; First posted 2019-10-16 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- No exercise control (Other): The investigators will use a randomised, crossover design study, where all subjects will complete (i) no exercise; (ii) 175kcal exercise; (iii) 350kcal exercise; and (iv) 700kcal exercise on a cycle ergometer the day before an oral glucose tolerance test (OGTT).
  350kcal has previously been shown to improve control of blood glucose when an OGTT is competed 24 h after the cycle ergometry exercise. The investigators have therefore chosen half this amount (175kcal) and double this amount (700kcal) to try and stimulate the greatest (700kcal) and least (175kcal) improvements in glycaemic control compared to no exercise. The investigators are, in essence, calculating a dose-response curve for quantity of exercise ((i) no exercise; (ii) 175kcal exercise; (iii) 350kcal exercise; and (iv) 700kcal exercise on a cycle ergometer) on the x axis and improvement in glycaemic control on the y axis.
  Interventions: Other: Cycle ergometry exercise at 60% VO2max
- 175kcal Cycle ergometry exercise at 60% VO2max (Experimental): The investigators will use a randomised, crossover design study, where all subjects will complete (i) no exercise; (ii) 175kcal exercise; (iii) 350kcal exercise; and (iv) 700kcal exercise on a cycle ergometer the day before an oral glucose tolerance test (OGTT).
  350kcal has previously been shown to improve control of blood glucose when an OGTT is competed 24 h after the cycle ergometry exercise. The investigators have therefore chosen half this amount (175kcal) and double this amount (700kcal) to try and stimulate the greatest (700kcal) and least (175kcal) improvements in glycaemic control compared to no exercise. The investigators are, in essence, calculating a dose-response curve for quantity of exercise ((i) no exercise; (ii) 175kcal exercise; (iii) 350kcal exercise; and (iv) 700kcal exercise on a cycle ergometer) on the x axis and improvement in glycaemic control on the y axis.
  Interventions: Other: Cycle ergometry exercise at 60% VO2max
- 350kcal Cycle ergometry exercise at 60% VO2max (Experimental): The investigators will use a randomised, crossover design study, where all subjects will complete (i) no exercise; (ii) 175kcal exercise; (iii) 350kcal exercise; and (iv) 700kcal exercise on a cycle ergometer the day before an oral glucose tolerance test (OGTT).
  350kcal has previously been shown to improve control of blood glucose when an OGTT is competed 24 h after the cycle ergometry exercise. The investigators have therefore chosen half this amount (175kcal) and double this amount (700kcal) to try and stimulate the greatest (700kcal) and least (175kcal) improvements in glycaemic control compared to no exercise. The investigators are, in essence, calculating a dose-response curve for quantity of exercise ((i) no exercise; (ii) 175kcal exercise; (iii) 350kcal exercise; and (iv) 700kcal exercise on a cycle ergometer) on the x axis and improvement in glycaemic control on the y axis.
  Interventions: Other: Cycle ergometry exercise at 60% VO2max
- 700kcal Cycle ergometry exercise at 60% VO2max (Experimental): The investigators will use a randomised, crossover design study, where all subjects will complete (i) no exercise; (ii) 175kcal exercise; (iii) 350kcal exercise; and (iv) 700kcal exercise on a cycle ergometer the day before an oral glucose tolerance test (OGTT).
  350kcal has previously been shown to improve control of blood glucose when an OGTT is competed 24 h after the cycle ergometry exercise. The investigators have therefore chosen half this amount (175kcal) and double this amount (700kcal) to try and stimulate the greatest (700kcal) and least (175kcal) improvements in glycaemic control compared to no exercise. The investigators are, in essence, calculating a dose-response curve for quantity of exercise ((i) no exercise; (ii) 175kcal exercise; (iii) 350kcal exercise; and (iv) 700kcal exercise on a cycle ergometer) on the x axis and improvement in glycaemic control on the y axis.
  Interventions: Other: Cycle ergometry exercise at 60% VO2max

INTERVENTIONS:
Other: Cycle ergometry exercise at 60% VO2max — Participants visit the lab on four occasions to complete (i) no exercise; (ii) 175kcal exercise; (iii) 350kcal exercise; (iv) or 700kcal exercise (randomised).

SUMMARY:
In 2015, there were 415 million adults worldwide with type II diabetes and by 2040, typeII diabetes will affect one in ten adults worldwide. Type II diabetes reduces quality of life and total lifespan, and two of the best countermeasures to type II diabetes are not drugs, but diet and exercise. Several studies have investigated the effects of exercise modality (aerobic, resistance, or concurrent) on glycaemic control and the mechanisms of these benefits. However, the minimal 'dose' of exercise required to increase insulin sensitivity and improve glycaemic control has never been established. Secondly, there is a progressive loss of muscle structure and function with age, which is known as sarcopenia. This study will also investigate whether the minimal amount of exercise is influenced by biological age and muscle mass by comparing physiological and biochemical responses in BMI-matched young and old volunteers. This study will therefore provide pilot data on the effect of age on exercise-mediated glycaemic control.

DETAILED DESCRIPTION:
Background Information and rationale Overarching aim: The purpose of this study is to identify the minimum number of calories that must be expended to improve the control of blood glucose in young and older overweight males, and in those with type II diabetes.

Why is this important? In 2015, there were 415 million adults worldwide with type II diabetes and by 2040, type II diabetes will affect one in ten adults worldwide. If the minimal volume of exercise to improve glycaemic control can be established, this could increase exercise compliance and population health.

Current knowledge and preliminary data Acute exercise improves glycaemic control by promoting the translocation of the glucose transporter GLUT-4 in an insulin-independent pathway. This mechanism is intact even in patients with type II diabetes. An acute bout of exercise for ~70 mins at 65% VO2max (energy expenditure of 350kcal) improves insulin sensitivity by ~15% 1h after exercise, and ~30% the day following exercise in obese adults. This improved insulin sensitivity is also associated with a 17% reduction in circulating free fatty acids, which chronically might benefit both type II diabetes and cardiovascular disease - a major secondary complication of type II diabetes. Several studies have investigated the effects of exercise modality (aerobic, resistance, or concurrent) on glycaemic control and the mechanisms of these benefits (8). However, the minimal 'dose' of exercise required to increase insulin sensitivity and improve glycaemic control has never been established. Secondly, there is a progressive loss of muscle structure and function with age, which is known as sarcopenia. This study will also investigate whether the minimal amount of exercise is influenced by biological age and muscle mass by comparing physiological and biochemical responses in BMI-matched young and old volunteers. Establishing the dose-response relationship for exercise and glycaemic control. It is important to establish the optimal dose-response relationship for exercise and glycaemic control in order to maximise the health benefits and minimize side-effects of the exercise intervention. Whilst the risks of exercise are low unless undertaking athlete-level training for several years, establishing the minimum exercise required for glycaemic control would improve exercise adherence. Indeed, lower volumes of exercise are easier to maintain than larger volumes, and this has led to the adoption of short-duration exercise strategies for glycaemic control, such as high intensity interval training.

Previous work has shown that an acute bout of cycling expending 350kcal can increase insulin sensitivity by ~30% the day following exercise in obese adults. On this basis, the proposed study will test three levels of kcal expenditure: 1) a 350kcal intervention, which is predicted to increase insulin sensitivity in line with; 2) a 700kcal intervention, to deliver a profound (doubling) stimulus to increase insulin sensitivity; and 3) 175kcal intervention, to examine the efficacy of a halved stimulus on insulin sensitivity. These three intervention points are necessary in order to accurately model the dose response relationship between amount of exercise and insulin sensitivity, which is currently unknown. There will also be a no exercise trial where the same data are collected and used to calculate baseline glycaemic control/insulin sensitivity from which any increase prompted by exercise can be determined. If the minimal volume of exercise to improve glycaemic control can be established, this could increase exercise compliance and population health. This minimal amount of exercise may increase in older subjects where muscle mass and quality is reduced. This study will therefore provide pilot data on the effect of age on exercise-mediated glycaemic control.

Objectives of the study Recruitment and testing will take place throughout the first 15 months of the study, allowing 3 months at the end of the study for data analysis. The investigators will use a randomised, crossover design study, where all subjects will complete (i) no exercise; (ii) 175kcal exercise; (iii) 350kcal exercise; and (iv) 700kcal exercise trials the day before an oral glucose tolerance test (OGTT). An acute bout of 350kcal exercise can improve insulin sensitivity by ~30% the following day; the trials in the proposed study intend to result in: (i) baseline glycaemic control; (ii) small improvements in glycaemic control; (iii) ~30% improvement in glycaemic control; and (iv) large >30% improvement in glycaemic control. The OGTT, continuous glucose monitoring (CGM), measurement of insulin, and FFA will be used to calculate dose response curves in each of these individual variables, where the minimum amount of exercise to improve glycaemic control can be ascertained.

ELIGIBILITY:
Cohort 1: 9 patients with type II diabetes under the following criteria:

Inclusion criteria

1. Aged 18 years and upwards
2. Capacity to consent to participation
3. Diagnosis of type II diabetes
4. BMI >25

Exclusion criteria

1. Patient is aged under 18 years
2. Patient lacks capacity to consent to participation
3. Anything that investigators feel affects the study measurements or safety

Cohort 2: 9 young control subjects under the following criteria:

Inclusion criteria

1. Aged 18 - 40
2. Capacity to consent to participation
3. BMI >25

Exclusion criteria

1. Subject is aged under 18 years
2. Subject lacks capacity to consent to participation
3. Subject on medication that affects glycaemic control
4. Anything that investigators feel affects the study measurements or safety

Cohort 3: 9 older control subjects under the following criteria:

Inclusion criteria

1. Aged >60
2. Capacity to consent to participation
3. BMI >25

Exclusion criteria

1. Subject is aged under 18 years
2. Subject lacks capacity to consent to participation
3. Subject on medication that affects glycaemic control
4. Anything that investigators feel affects the study measurements or safety

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-09-26 (Actual); Study Completion 2022-09-29 (Actual)

PRIMARY OUTCOMES:
Lowering of blood glucose values throughout the two-hour oral glucose tolerance test (OGTT) measured every 30 minutes throughout from an arterialised-venous hand vein 24 hours following large (700kcal) in comparison to small (175kcal) exercise quantities | over the 8 weeks of participant involvement in study
  The investigators will quantify the lowering of blood glucose values during the OGTT 24h following 175kcal, 350kcal and 700kcal exercise when compared to a no exercise control.

SECONDARY OUTCOMES:
Lowering of serum insulin values throughout the two-hour oral glucose tolerance test (OGTT) measured every 30 minutes throughout from an arterialised-venous hand vein 24 hours following large (700kcal) in comparison to small (175kcal) exercise quantities | over the 8 weeks of participant involvement in study
  The investigators will quantify the lowering of serum insulin values during the OGTT 24h following 175kcal, 350kcal and 700kcal exercise when compared to a no exercise control.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Lancaster Infirmary, Lancaster, United Kingdom

IPD SHARING:
Plan to Share IPD: No